CLINICAL TRIAL: NCT05599321
Title: Piloting a Virtual Navigation (VN) System for Bronchoscopic Lung Nodule Sampling
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, William E. Higgins, Distinguished Professor, Penn State University
Other Study IDs: 20714
Record Dates: First submitted 2022-10-13; First posted 2022-10-31 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: bronchoscopy; computer-assisted surgery; image-guided surgery; surgical navigation; image-guided biopsy; multimodal imaging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical Controls Cohort: Lung cancer patients who have previously undergone a clinical bronchoscopy. This group represents the current state-of-the-art bronchoscopy practice.
- Consented Clinical Bronchoscopy Cohort: Lung cancer patients, scheduled for bronchoscopy, who are consented for bronchoscopy assisted by the Virtual Navigator.
  Interventions: Diagnostic Test: Virtual Navigation System

INTERVENTIONS:
Diagnostic Test: Virtual Navigation System — The Virtual Navigator guidance computer is interfaced to the bronchoscopy hardware to tap off the live bronchoscopy and EBUS video feeds. The standard OR medical team (technicians, clinical fellows, et al.) is on hand, and standard clinical facilities (e.g., fluoroscopy, CT/PET image viewer) are available. Our technical team is also present to record all procedural video and computer display information. It also operates the guidance computer during the guided procedure and offers any assistance in case of unanticipated issues. The participant's clinical bronchoscopy will be recorded by the radiology imaging management system.
  Groups: Consented Clinical Bronchoscopy Cohort

SUMMARY:
The overall goal is to evaluate the role of a Virtual Navigation (VN) system (the Virtual Navigator) in the bronchoscopic evaluation and tissue sampling of lung cancer and other chest lesions at the Penn State Hershey Medical Center (HMC). The Virtual Navigator is a software package that runs on a mobile Windows-based computer. The computer takes in up to four clinical image/video sources, ordered by the clinician for clinical purposes: 1) 3D CT (computed tomography) imaging scan; 2) 3D PET (positron emission tomography) imaging scan (optional); 3) Bronchoscopic video of the airway tree interior; 4) Ultrasound video of scanned anatomy outside the airways, as provided by an endobronchial ultrasound (EBUS) probe (optional). During a live guided procedure, the Virtual Navigator presents images that assist with navigating the bronchoscope to predesignated chest lesions.

Lung cancer patients that present a suspicious peripheral tumor on their chest CT scan are often prescribed to undergo a diagnosis-and-staging bronchoscopy, whereby the bronchoscopist examines both the suspect tumor and any identified central-chest lymph nodes. For the clinical study, we consider bronchoscopy performance for two cohorts: 1) a cohort of consented patients who undergo image-guided bronchoscopy via the Virtual Navigator; and 2) a historical controls cohort consisting of patients who underwent bronchoscopy recently at our medical center (state-of-the-art bronchoscopy practice). The study's general hypothesis is that an image-guided bronchoscopy system (the Virtual Navigator) that integrates 3D imaging, bronchoscopy, and EBUS images enables more complete evaluation and sampling of chest lesions than current state-of-the-art clinical techniques. More specifically, for peripheral-tumor diagnosis, the sub-hypothesis is that the VN system increases diagnostic biopsy yield as compared to state-of-the-art bronchoscopy practice; for central-chest nodal staging, the sub-hypothesis is that the VN system enables the sampling of more lymph nodes than state-of-the-art bronchoscopy practice.

ELIGIBILITY:
Inclusion Criteria:

* patients from age 18 and over
* a planned clinical bronchoscopy to evaluate abnormal lung parenchyma and/or central chest lymph nodes
* a clinical CT scan performed at Hershey Medical Center that meets technical specifications and is available on the Radiology research server
* (Optional, use if available) CT/PET images that meet technical specifications and are available on the Hershey Medical Center clinical image storage system

Exclusion Criteria:

* inability to give consent
* the CT scan does not meet technical specifications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population includes patients whose clinical evaluation requires a diagnostic bronchoscopy for evaluation of parenchymal or mediastinal abnormalities. This patient population is typically 40-70 years old.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety measurement | 1 years
  Presence or absence of errors in the VN System during bronchoscopic procedure
Functionality measurement | 1 years
  Presence or absence of software malfunctions in the VN System during bronchoscopic procedure
Diagnostic biopsy yield | 2 years
  Comparison of diagnostic biopsy yield between the live cases and historical controls
Number of lymph nodes visited | 2 years
  Comparison of number of lymph nodes visited between the live cases and historical controls

SECONDARY OUTCOMES:
Biopsy samples | 2 years
  Number of biopsy samples taken per tumor or lymph node
Tumor pathology | 2 years
  Whether a sample is malignant, non-malignant, or indeterminate and adequacy of sample
Procedure complications | 2 years
  Rate of complications from bronchoscopic procedure
Distance from biopsy site to optimal site | 2 years
  Distance between actual biopsy site and computed optimal biopsy site
Procedure time | 2 years
  Procedure time (total and per tumor or lymph node) in minutes

CONTACTS AND LOCATIONS:
Overall Officials: William E Higgins, PhD, Principal Investigator — Penn State University, University Park, PA 16802; Rebecca Bascom, MD, Study Director — Penn State Milton S. Hershey Medical Center, Hershey, PA 17033
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States